CLINICAL TRIAL: NCT03058562
Title: A Randomized, Placebo-Controlled, Single-Dose Crossover Study of ABX-1431 HCl in Adult Patients With Tourette Syndrome (TS) and Chronic Motor Tic Disorder
Brief Title: A Study to Evaluate the Effects of ABX-1431 on Patients With Tourette Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abide Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: ABX-1431_PN015
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Tourette Syndrome; Chronic Motor Tic Disorder
MeSH Terms: conditions — Tourette Syndrome | interventions — ABX-1431

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Crossover Sequence A (Experimental): Each in the fasting state:
  Period 1: Single-dose matching placebo
  Period 2: Single-dose ABX-1431
  Interventions: Drug: ABX-1431; Drug: Placebo Comparator
- Crossover Sequence B (Experimental): Each in the fasting state:
  Period 1: Single-dose ABX-1431
  Period 2: Single-dose matching placebo
  Interventions: Drug: ABX-1431; Drug: Placebo Comparator
- Crossover Sequence C (Experimental): Each with a standard high fat meal:
  Period 3: Single-dose matching placebo
  Period 4: Single-dose ABX-1431
  Interventions: Drug: Placebo Comparator; Drug: ABX-1431
- Crossover Sequence D (Experimental): Each with a standard high fat meal:
  Period 3: Single-dose ABX-1431
  Period 4: Single-dose matching placebo
  Interventions: Drug: Placebo Comparator; Drug: ABX-1431

INTERVENTIONS:
Drug: ABX-1431 — ABX-1431, capsules, 40 mg in the fasting state
  Arms: Crossover Sequence A; Crossover Sequence B
Drug: Placebo Comparator — Matching Placebo
Drug: ABX-1431 — ABX-1431, capsules, 20 mg with a high fat meal
  Arms: Crossover Sequence C; Crossover Sequence D

SUMMARY:
The study will investigate the effects and the safety of a single-dose of ABX-1431 HCl on tics and other symptoms of Tourette Syndrome.

During part 1 (periods 1 and 2) each patient will receive study drug once and placebo once.

Patients who complete part 1 with adequate clinical safety will be offered the option to participate in part 2 (periods 3 and 4) and again willl receive study drug once and placebo once where, in contrast to part 1, administration will take place with a standard high fat meal.

DETAILED DESCRIPTION:
This is a single dose, double-blind, randomized, placebo-controlled, cross-over study. This study will assess the single dose effects of ABX-1431 HCl on tics and other symptoms of Tourette Syndrome.

All patients will undergo a screening visit for enrollment criteria. Eligible patients will be treated with a single dose of ABX-1431 HCl or placebo followed by efficacy, safety and pharmacokinetics assessments. After a washout period of 1-3 weeks, patients will undergo identical procedures with the other treatment.

Only patients who complete the first part of the study with adequate clinical safety will be offered the option to participate in an additional two period crossover, where ABX-1431 HCl or placebo is taken with a standard high fat meal. Again, efficacy, safety and pharmacokinetics assessments will be done. After a washout period of 1-3 weeks, patients will undergo identical procedures with the other treatment.

This study will enroll 20 patients with a diagnosis of Tourette Syndrome OR chronic motor tic disorder.

ELIGIBILITY:
Principal Inclusion Criteria:

* Patient is a male or female between the age of 18 and 65 years of age at the Screening Visit.
* Patient has a diagnosis of Tourette Syndrome OR chronic motor tic disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria.
* Patient's Yale Global Tic Severity Scale (YGTSS) total tic sub-scale (TTS) results must be ≥ 18 (Range 0-50) at the Screening Visit.
* Patients taking daily medications for symptoms of Tourette Syndrome [e.g. neuroleptics (e.g. aripiprazole, risperidone) or selective serotonin reuptake inhibitors (e.g. fluoxetine)] must be on a stable dose of medication for at least 30 days before the Screening Visit and must be expected to remain on a stable dose during this study.

Principal Exclusion Criteria:

* Patient is taking potent cytochrome P450 3A4/5 inducers [e.g. carbamazepine, oxcarbazine, rifampin, St. John's Wort (Hypericum perforatum), or phenytoin]. Patient is taking strong P450 3A4/5 inhibitors including atazanavir, bocepravir, clarithromycin, grapefruit juice, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telithromycin, or voriconazole.
* Patients with a diagnosis of any psychiatric comorbidity (obsessive compulsive disorder, attention deficit hyperactivity disorder) OR generalized anxiety disorder, depression or post-traumatic stress disorder that is unstable or requires alteration in therapy are excluded. Patients with a past history of psychosis or schizophrenia at any time are excluded. Patients with stable OCD or ADHD requiring no alteration in therapy may be enrolled.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-10-04 (Actual); Study Completion 2017-10-04 (Actual)

PRIMARY OUTCOMES:
Change of rating in Modified Rush Video Scale (MRVS) over time | pre-dose, post-dose (4 hours, 8 hours)
Change in rating of Yale Global Tic Severity Scale (YGTSS) over time | pre-dose, post-dose (4 hours, 8 hours)
Change of rating in Adult Tic Questionnaire (ATQ) over time | pre-dose, post-dose (4 hours, 8 hours, 12 hours)
Change of rating in Premonitory Urge for Tics Scale (PUTS) over time | pre-dose, post-dose (4 hours, 8 hours, 12 hours)

SECONDARY OUTCOMES:
ABX-1431 and metabolite (M55) plasma pharmacokinetics | pre-dose, post-dose (2 hours, 4 hours, 8 hours, 24 hours)
2-AG hydrolysis in PBMC | pre-dose, post-dose (2 hours, 4 hours, 8 hours, 24 hours)
Number and severity of adverse events (AEs), serious adverse events (SAEs), and suspected unexpected serious adverse reactions (SUSARs) | screening, pre-dose, post-dose (0 hours, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours), follow-up
Number of patients with clinically significant change in vital signs | screening, pre-dose, post-dose (2 hours, 4 hours, 8 hours, 24 hours)
  The following vital signs will be assessed:
  heart rate, blood pressure, respiratory rate, temperature
Number of patients with clinically significant change in Laboratory safety tests | screening, pre-dose, post-dose (24 hours)
  The following laboratory safety tests will be assessed:
  Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Albumin, Alkaline phosphatase, Bicarbonate, Calcium, Chloride, Cholesterol, Creatinine, Glucose, Potassium, Sodium, Bilirubin, total (bilirubin to be fractionated if total bilirubin is elevated), Blood urea nitrogen (BUN)/Urea, hemoglobin, hematocrit, red blood cell (RBC) count, platelet count, white blood cell (WBC) count (total and differential count), polymorphonuclear leukocytes (neutrophils), lymphocytes, eosinophils, monocytes, basophils; Urinalysis: pH, specific gravity, glucose, ketones, leukocyte, esterase, nitrites, occult blood, protein
12-lead ECG assessments | screening, pre-dose, post-dose (4 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Chan Beals, Study Director — Abide Therapeutics, Inc.
Locations (1):
- Medizinische Hochschule Hannover, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No